CLINICAL TRIAL: NCT03794674
Title: Validation of a Record-based Frailty Assessment According to the Multidimensional Prognostic Index
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: MPIRECVALID
Record Dates: First submitted 2018-12-21; First posted 2019-01-07 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2018-12

CONDITIONS: Frail Elderly Syndrome
Keywords: Multidimensional Prognostic Index; Frailty; Geriatric; Elderly; Aged; +75; Comprehensive Geriatric Assessment
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MPI test group: 50 eligible patients. Frailty level independently assessed by two reviewers based on the medical records and assessed by one research assistant based on bedside testing.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — No intervention, since this is a validation study

SUMMARY:
Background Various phenotype and cumulative frailty assessment tools have been developed and compared in research. For use in an in-hospital setting, a cumulative and graded frailty assessment method is preferred in order to identify subgroups of patients at risk of adverse events during discharge and transition to primary care. Comprehensive Geriatric Assessment (CGA) is the gold standard to assess frailty. Most medical wards have limited access to specialized geriatric team support capable of performing CGA. Thus in these wards there is a need for a CGA based instrument to identify the frail patients and to quantify the level of frailty. The Multidimensional Prognostic Index (MPI) is based on CGA and is a comprehensive cumulative deficit frailty assessment tool validated in a Danish geriatric department. MPI is fully applicable in the everyday clinical work and supplies useful information to clinicians. It can predict readmission and death, and it is well-suited to assess the degree of frailty. Enabling identification of patients at risk of adverse events facilitates targeting of the interventions in order to improve patient outcomes. The MPI is a bedside assessment. However, in observational record-based research the patient is not accessible for the researcher. To assess and identify hospitalized frail patients retrospectively for clinical research, a valid record-based frailty assessment method is needed. The aim of this study is to compare the accuracy of a record-based MPI assessment with a bedside performed MPI assessment in order to use the record-based MPI when access to bedside MPI is impossible.

ELIGIBILITY:
Inclusion Criteria:

* Acutely admitted to one of the two medical departments listed below
* Aged 75 years or older
* Living within the municipality of Aarhus

Exclusion Criteria:

* Included in any other kind of follow-up schemes
* Already included in this study
* Declared terminally ill or undergoing palliative care at admission
* Admitted from one specific temporary nursing home with geriatric medical assistance (Vikærgården)
* Discharge or transfer to another department, including hospice
* The patient does not want to participate in the MPI-screening process

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study group comprises medical patients acutely admitted to the Department of Cardiology and the Department of Infectious Diseases, Aarhus University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Sumscore | 1 day
  The relative difference between the two measurements' sumscores calculated as an Intraclass Correlation Coefficient (ICC)

CONTACTS AND LOCATIONS:
Overall Officials: Troels Hansen, MD, Principal Investigator — Aarhus University Hospital and Aarhus University
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dent E, Kowal P, Hoogendijk EO. Frailty measurement in research and clinical practice: A review. Eur J Intern Med. 2016 Jun;31:3-10. doi: 10.1016/j.ejim.2016.03.007. Epub 2016 Mar 31. PMID 27039014
- [Background] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Background] Volpato S, Bazzano S, Fontana A, Ferrucci L, Pilotto A; MPI-TriVeneto Study Group. Multidimensional Prognostic Index predicts mortality and length of stay during hospitalization in the older patients: a multicenter prospective study. J Gerontol A Biol Sci Med Sci. 2015 Mar;70(3):325-31. doi: 10.1093/gerona/glu167. Epub 2014 Sep 9. PMID 25209253
- [Background] Pilotto A, Ferrucci L, Franceschi M, D'Ambrosio LP, Scarcelli C, Cascavilla L, Paris F, Placentino G, Seripa D, Dallapiccola B, Leandro G. Development and validation of a multidimensional prognostic index for one-year mortality from comprehensive geriatric assessment in hospitalized older patients. Rejuvenation Res. 2008 Feb;11(1):151-61. doi: 10.1089/rej.2007.0569. PMID 18173367
- [Background] Gregersen M, Hansen TK, Jørgensen BB, Damsgaard EM. Validation of a modified Multidimensional Prognostic Index obtained at discharge in older Danish geriatric patients to predict acute readmission and mortality. 2018 Unpublished data.
- [Background] Warnier RM, van Rossum E, van Velthuijsen E, Mulder WJ, Schols JM, Kempen GI. Validity, Reliability and Feasibility of Tools to Identify Frail Older Patients in Inpatient Hospital Care: A Systematic Review. J Nutr Health Aging. 2016 Feb;20(2):218-30. doi: 10.1007/s12603-015-0567-z. PMID 26812520
- [Background] Hopkins WG. Measures of reliability in sports medicine and science. Sports Med. 2000 Jul;30(1):1-15. doi: 10.2165/00007256-200030010-00001. PMID 10907753
- [Background] de Vet HC, Terwee CB, Knol DL, Bouter LM. When to use agreement versus reliability measures. J Clin Epidemiol. 2006 Oct;59(10):1033-9. doi: 10.1016/j.jclinepi.2005.10.015. Epub 2006 Aug 10. PMID 16980142
- [Background] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT03794674/Prot_SAP_001.pdf